CLINICAL TRIAL: NCT00086424
Title: Epidemiology of Insulin Growth Factor (IGF) and Cardiovascular Events
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Robert Kaplan, Prof. Epidemiology & Population Health, Albert Einstein College of Medicine
Other Study IDs: 1259; 5R01HL075516 (NIH); 1R01AG031890 (NIH); 2003-020 (Other: Albert Einstein College of Medicine-IRB)
Record Dates: First submitted 2004-07-01; First posted 2004-07-05 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Cerebrovascular Accident; Heart Failure; Heart Failure, Congestive
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Stroke; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the role of insulin growth factor in cardiovascular disease in older men and women.

DETAILED DESCRIPTION:
BACKGROUND:

Insulin-like growth factor-I (IGF-I) is the main mediator of effects of growth hormone (GH) and an important regulator of cell cycle/differentiation and inhibitor of apoptosis. Consistent with laboratory studies showing potentially beneficial effects of IGF-I on the cardiovascular and cerebrovascular systems, GH-deficient individuals have high cardiovascular disease (CVD) mortality and evidence of premature atherosclerotic disease that is reversible with GH replacement. In addition, several epidemiological and clinical studies have shown an association between low serum IGF-I levels and myocardial infarction (MI) and congestive heart failure (CHF) among persons without frank abnormalities of the GH/IGF-I axis.

DESIGN NARRATIVE:

The study is the first prospective investigation to assess whether serum levels of IGF-I and two of its important binding proteins, IGFBP-3, and IGFBP-1, are associated with incidence of confirmed incident cardiovascular disease (CVD) events in older male and female adults. Specimens and data for this study will be obtained from the Cardiovascular Health Study (CHS), a large, multi-center NHLBI-funded prospective cohort study of 5,888 community-dwelling men and women 65 years or older. The study uses an efficient case-cohort study design to select specimens for testing, involving evaluation of 750 incident myocardial infarction (MI)/fatal coronary heart disease (CHD) cases, 500 incident stroke cases, 750 incident congestive heart failure (CHF) cases, and a comparison sub-cohort of 750 individuals selected at random from the study population. The study examines the association between baseline serum IGF-I, IGFBP-1, and IGFBP-3 level and the future occurrence of first incident MI/fatal CHD, ischemic stroke, and CHF. Multivariate regression models are used to control for potential confounding factors including age, sex, race/ethnicity, anthropometry and body composition, fasting and 2-hour post-load glucose and insulin levels, dietary intake, physical activity, hormone replacement therapy and other medications, and other CVD risk markers such as lipids, inflammatory factors, and coagulation/fibrinolysis markers.

ELIGIBILITY:
Medicare-eligible adults as well as other age-eligible individuals residing in the household

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community dwelling adults aged 65 years and older recruited from four US field centers
Sampling Method: Probability Sample
Enrollment: 5888 (Actual)
Dates: Start 2004-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Kaplan, Ph.D., Principal Investigator — Albert Einstein College of Medicine